CLINICAL TRIAL: NCT01404013
Title: Randomised, Open-label, Parallel-group Study of Therapeutic Effect of Leukotriene Modulator Montelukast Alone or Combined With Inhaled Corticosteroid on Cough Variant Asthma
Brief Title: Effects of Leukotriene Modulator Montelukast on Cough Variant Asthma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Kefang Lai, professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MISP 39227
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2012-11

CONDITIONS: Asthma
Keywords: Montelukast; Cough variant asthma; Inhaled Corticosteroid
MeSH Terms: conditions — Asthma; Cough-Variant Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Montelukast (Active Comparator): Monotherapy with Montelukast 10mg, take orally ,every night,for 8 weeks
  Interventions: Drug: Montelukast
- ICS/LABA and Montelukast (Active Comparator): Combination therapy with inhaled corticosteroid/β2 agonist 160/4.5ug,twice a day and Montelukast 10mg，take orally,every night for 8 weeks
  Interventions: Drug: ICS/LABA and Montelukast
- ICS/LABA (Active Comparator): Monotherapy with corticosteroid/β2 agonist 160/4.5ug,inhaled, twice a day, for 8 weeks
  Interventions: Drug: ICS/LABA

INTERVENTIONS:
Drug: ICS/LABA — Budesonide 160µg and Formoterol 4.5µg, 1puff ,twice a day, for 8 weeks
  Other Names: Symbicort Turbuhaler
  Arms: ICS/LABA
Drug: Montelukast — Montelukast 10mg ,every night, for 8 weeks
  Other Names: Singulair
  Arms: Montelukast
Drug: ICS/LABA and Montelukast — Budesonide 160µg and Formoterol 4.5µg, 1puff, twice a day, for 8 weeks; Montelukast 10mg ,take orally ,every night for 8 weeks
  Other Names: Inhaled corticosteroid/β2 agonist: Symbicort Turbuhaler; Montelukast: Singulair
  Arms: ICS/LABA and Montelukast

SUMMARY:
This study aims to observe the therapeutic effect of leukotriene modulator montelukast alone or combined with inhaled corticosteroid(ICS) on cough variant asthma(CVA).

The investigators hypothesize:

1. Cough score and cough reflex sensitivity will be improved after treatment with montelukast, inhaled corticosteroid/β2 agonist(ICS/LABA), and two combinations.
2. Combination of leukotriene modulator and inhaled corticosteroid/β2 agonist may have better efficacy when compared to montelukast, corticosteroid/β2 agonist alone while MON, is comparable to symbicort.

DETAILED DESCRIPTION:
Study groups:

99 patients diagnosed with CVA will be randomised into three groups as follows:

Group 1: inhaled corticosteroid+β2 agonist The patients with cough variant asthma received Symbicort Turbuhaler (Budesonide 160µg and Formoterol 4.5µg) 1puff Q12h for 8 weeks.

Group 2: montelukast The patients with cough variant asthma received montelukast 10mg QN for 8 weeks, without any other corticosteroid or β2 agonist.

Group 3: montelukast combined with inhaled corticosteroid+β2 agonist The patients with cough variant asthma received montelukast 10mg QN combined with Symbicort Turbuhaler (Budesonide 160µg and Formoterol 4.5µg) 1puff Q12h for 8 weeks..

The study will be divided into following phases:

1. First Visit (Visit 1, day -6):

   A full medical history and physical examination to be undertaken to determine whether patients meet the inclusion/exclusion criteria.

   After the informed consent has been signed, the following samples are obtained from all patients: blood samples for routine clinical laboratory tests (haematology, biochemistry and chest x-ray). A urine pregnancy test will be performed in women of childbearing potential.

   Bronchial provocation test by methacholine inhalation are performed to determined the presence of bronchial non-specific hyper-responsiveness.

   Patients are given the Diary Card.
2. Screening Period ( day -6 to day 0, 6 Days) Patients took two medications as bellows for 3 days and followed by 3 days of wash-out period. Patients should completed 6 days diary card, starting from day -6 to week 0.

   Bambuterol HCI (Bambec, brand name), 10 mg qn po Theophylline tablet sustained release, 100mg bid po
3. Second Visit (Visit 2, Week 0):

   A physical examination were to be performed. All laboratory tests results are obtained to determine whether patients meet the inclusion/exclusion criteria. Concurrent medication were recorded.

   The Diary Card were collected, reviewed and assessed whether ICS, bronchodilator or ICS/BD treatment is efficient for cough symptom (symptom score improved 1 at least).

   Capsaicin challenge test and FENO were performed and hypertonic saline induced sputum samples for cell differential, urine leukotriene, serum IgE, were taken from enrolled patients.

   Enrolled patients were randomized into different groups, and the study medication were dispensed.
4. During Treatment 1(Week 0 to Week 4, 14 days):

   Patients were to take study medication for 28 days and completed Diary Card for 7 days from Week 3 to Week 4.
5. Third Visit (Visit 3, Week 4):

   A physical examination were to be performed. The Diary Card were collected and reviewed. Adverse events, secondary complications, concurrent medication will be recorded.

   Capsaicin challenge test and FENO were performed and hypertonic saline induced sputum samples for cell differential were taken from enrolled patients.
6. During Treatment 2 (Week 4 to Week 8, 14 days):

   Patients were to take study medication for 28 days and completed Diary Card for 7 days from Week 7 to Week 8.
7. Forth Visit (Visit 4, Week 8):

A physical examination and were to be performed. The Diary Card were collected and reviewed. Residual (unused) medications were to be returned. Adverse events, secondary complications, concurrent medication will be recorded.

Capsaicin challenge test and FENO were performed and hypertonic saline induced sputum samples for cell differential, urine leukotriene, serum IgE, were taken from enrolled patients.

Blood samples for routine clinical laboratory tests (haematology and biochemistry) were obtained, if a clinically significant laboratory abnormal result was noted at the visit 4, AE and a follow-up visit would be considered.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have a history of cough as sole or main symptom lasting more than 8 weeks, often irritating cough more cough at night.
2. Patients who were diagnosed with positive result in bronchial provocation test by methacholine inhalation challenge.
3. There is evidence that bronchodilator treatment* is efficient for cough symptom (symptom score improved 1 at least).
4. Patients whose chest x-ray outcome was normal or without any active focus.
5. Patients who was aged from 18 years old (≥ 18 years old ) to 75 years old (≤ 75 years old).

Exclusion Criteria:

1. Patients demonstrate FEV1/FVC <70% in lung function test. FEV1 stands for forced expiratory volume in 1 second, FVC stands for forced vital capacity.
2. Patients who is a smoker or ex-smoker and has smoked within the previous year or has a cumulative smoking history >10 pack-years or equivalence.
3. Patients with concomitance of GERC (gastroesophageal reflux-related chronic cough), chronic bronchitis , bronchiectasis, bronchial tuberculosis, ACEI induced cough, bronchogenic carcinoma, psychologic cough, pulmonary fibrosis, bronchus foreign body, microlithiasis, tracheobroncheopathia osteochondroplastica, mediastinal tumor, left ventricular dysfunction.
4. Female subjects who are pregnant, breast-feeding or risk of becoming pregnant during the study.
5. Subjects who are known or suspected to be hypersensitive to any component of the study medication or relief medications.
6. Subjects who have received any therapy in the previous seven days, e.g. oral/ inhaled/systematic corticosteroid, long-acting β2 agonist, theophylline sustained release.
7. Subjects who are diagnosed with past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, endocrine disease or pulmonary disease. e.g.nasal-sinus infection, lower respiratory tract infection, chronic bronchitis, emphysema, bronchiectasis, cystic fibrosis or bronchopulmonary dysplasia.
8. Subjects who demonstrate significant abnormality on biochemistry, hematology, ECG.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Day-time and night-time cough symptom total-score changes from baseline to visit 4 | 8 weeks

SECONDARY OUTCOMES:
Cough reflex sensitivity changes in different groups at baseline, visit 2, visit3, and visit 4. Cell differential changes in hypertonic saline induced sputum in different groups at baseline, visit 2, visit3, and visit 4. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mengfeng Li, MD., Study Chair — Sun Yat-sen University
Locations (1):
- Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Yi F, Zhan C, Liu B, Li H, Zhou J, Tang J, Peng W, Luo W, Chen Q, Lai K. Effects of treatment with montelukast alone, budesonide/formoterol alone and a combination of both in cough variant asthma. Respir Res. 2022 Oct 10;23(1):279. doi: 10.1186/s12931-022-02114-6. PMID 36217131